

Zhejiang Teruisi Pharmaceutical Inc.

## Table/Figure/Listing Shells

A RANDOMIZED, DOUBLE-BLIND, SINGLE-DOSE, THREE-ARM, PARALLEL-GROUP, PHASE 1 STUDY TO COMPARE PHARMACOKINETIC AND SAFETY OF TRS003 TO CHINA-APPROVED BEVACIZUMAB AND US-LICENSED AVASTIN, WHEN ADMINISTERED INTRAVENOUSLY TO HEALTHY MALE SUBJECTS

Sponsor Study No. TRS00301001 inVentiv Health Clinique Inc. Project No. 182013

Final Version: 1.0 Date: 19-SEP-2018

Contract Research Organization: inVentiv Health Clinique Research Services LLC (inVentiv), a Syneos Health company 1951 NW 7th Avenue, Suite 450 Miami, FL 33136, USA Sponsor: Zhejiang Teruisi Pharmaceutical Inc. 1207, Building 3, 1366 Hongfeng Road,

Huzhou, Zhejiang, 313000 China

### **CONFIDENTIAL**



Zhejiang Teruisi Pharmaceutical Inc.

## **SIGNATURES**

Sponsor Study No.: TRS00301001

in Ventiv Project No.: 182013

Study Title: A Randomized, Double-Blind, Single-Dose, Three-Arm, Parallel-Group, Phase 1 Study to Compare Pharmacokinetic and Safety of TRS003 to China-Approved Bevacizumab and US-Licensed Avastin, When Administered Intravenously to Healthy Male Subjects.

Author:

Uttam Hubale, M. Sc.

Statistician inVentiv

Signature: Date:

Sponsor's

Representative: Dr Libin Zhao

Medical Monitor

Zhejiang Teruisi Pharmaceutical Inc.

Signature:

Date:



Zhejiang Teruisi Pharmaceutical Inc.

## TABLE OF CONTENTS

| SIG | GNATURES | 2 |
|-----|----------------------------------------------|----|
| TAI | BLE OF CONTENTS | 3 |
| 1. | Tables, Figures and Data Listings Formatting | 4 |
| | Table 1-1 Layout Specifications | |
| 2. | Summary TFLs | |
| | Table 2-1 List of Table Shells | |
| | Table 2-2 List of Figures Shells | 7 |
| | Table 2-3 List of Data Listings Shells | |
| 3. | CSR In-text Tables | 9 |
| 4. | Summary Tables | 14 |
| 5. | Figures | 40 |
| 6. | Listings | 47 |

Zhejiang Teruisi Pharmaceutical Inc.

## 1. Tables, Figures and Data Listings Formatting

The table, figure, and data listing (TFL) shells are presented in order to provide a framework for displaying the study data. The shells may change due to unforeseen circumstances. The shells may not be truly representative of every aspect of the study (e.g., sampling time points, assessed laboratory parameters, calculated parameters, units), but are intended to illustrate the general layout of the tables, figures, and data listings that will be included in the final report.

The default tables, listings, and figures layout will be as presented in Table 1-1:

**Table 1-1 Layout Specifications** 

| Orientation | Portrait | Landscape |
|---|---|---|
| Paper Size | Letter | Letter |
| Margins | Top: 3.05 cm | Top: 3.05 cm |
| | Bottom: 2.54 cm | Bottom: 2.2 cm |
| | Left: 2.54 cm | Left: 1.9 cm |
| | Right: 2.54 cm | Right: 1.9 cm |
| Font | Table text: Times new Ro | Table text: Times new Roman 9 or 10 pts |
| | Table title: Times new Ro | Table title: Times new Roman 12 pts |
| | Table legend: Times new | Roman 10 pts |

The font size may be reduced as necessary to allow additional columns to be presented, but not at the expense of clarity. Also the orientation may be changed to portrait if appropriate.

Except for pharmacokinetic (PK) tables, descriptive statistics for minimum and maximum will be presented with the same decimal digits as the original values, and with one more decimal place than the original data for mean, standard Deviation, and median. For PK tables, the data presentation will be as per the appropriate inVentiv SOP.



## 2. Summary TFLs

# **Table 2-1 List of Table Shells**

| Table<br>Number | Title |
|---|---|
| | In-Text Table |
| 10.1-1 | Subject Disposition |
| 11.4.2.3-1 | Summary of Pharmacokinetic Parameters – PK Population |
| 11.4.2.3-2 | Ratios (A/B and C/B), 90% Geometric Confidence Intervals, Inter-Subjects CV (%) and P-value – PK Population |
| 11.4.2.3-3 | Ratios (A/C), 90% Geometric Confidence Intervals, Inter-Subjects CV (%) and P-value – PK Population |
| | Demographic Data Summary Tables |
| 14.1-1 | Summary of Demographic Characteristics of Subjects Included in the Safety Population |
| 14.1-2 | Summary of Demographic Characteristics of Subjects Included in the Pharmacokinetic Population |
| | Pharmacokinetic Tables |
| 14.2.1-1 | Descriptive Statistics of Bevacizumab Plasma Concentration over Nominal Time by Treatment - PK Population |
| 14.2.1-2 | Descriptive Statistics of Bevacizumab Pharmacokinetic Parameters by Treatment - PK Population |
| 14.2.1-3 | Ratios (A/B, A/C and C/B), 90% Geometric Confidence Intervals, Inter-Subjects CV (%) and P-value – PK Population |
| | Safety Data Summary Tables |
| 14.3.1-1 | Frequency of Subjects Experiencing Treatment-Emergent Adverse Events and Number of Events Summarized per Treatment – Safety Population |
| 14.3.1-2 | Frequency of Subjects Experiencing Treatment-Emergent Adverse Events Summarized per Treatment and Severity – Safety Population |
| 14.3.1-3 | Number of Treatment-Emergent Adverse Events Summarized per Treatment and Severity – Safety Population |
| 14.3.1-4 | Frequency of Subjects Experiencing Treatment-Emergent Adverse Events Summarized per Treatment and Relationship – Safety Population |
| 14.3.1-5 | Number of Treatment-Emergent Adverse Events Summarized per Treatment and Relationship – Safety Population |
| 14.3.4-1 | Biochemistry Summary Descriptive Statistics – Safety Population |
| 14.3.4-2 | Frequency of Subjects – Biochemistry Shifts from Baseline – Safety Population |
| 14.3.4-3 | Hematology Summary Descriptive Statistics – Safety Population |
| 14.3.4-4 | Frequency of Subjects – Hematology Shifts from Baseline – Safety Population |
| 14.3.4-5 | Urinalysis (pH and Specific Gravity) Summary Descriptive Statistics – Safety Population |



Zhejiang Teruisi Pharmaceutical Inc.

| 14.3.4-6 | Frequency of Subjects – Urinalysis (pH and Specific Gravity) Shifts from Baseline – Safety Population |
|---|---|
| 14.3.4-7 | Urinalysis Frequency Summary - Categorical Results - Safety Population |
| | Frequency of Subjects – Urinalysis Shifts from Baseline – Categorical Results – Safety |
| 14.3.4-8 | Population |
| 14.3.4-9 | Vital Signs Summary Descriptive Statistics – Safety Population |
| 14.3.4-10 | Electrocardiogram Summary Descriptive Statistics – Safety Population |
| 14.3.4-11 | Descriptive Statistics of Immunogenicity - Safety Population |

Zhejiang Teruisi Pharmaceutical Inc.

## **Table 2-2 List of Figures Shells**

| Figure<br>Number* | Title |
|---|---|
| 14.2.2-1a to | Plasma Concentrations for Subject XX - Linear Scale |
| 14.2.2-114a** | |
| 14.2.2-1b to | Plasma Concentrations for Subject XX - Semi-Log Scale |
| 14.2.2-114b** | |
| 14.2.2-115a | Mean (± SD) Plasma Concentrations - Linear Scale |
| 14.2.2-115b | Mean (± SD) Plasma Concentrations - Semi-Log Scale |
| 14.2.2-116a | Overlay of Individual and Mean Plasma Concentrations by Treatment - Linear Scale |
| 14.2.2-116b | Overlay of Individual and Mean Plasma Concentrations by Treatment - Semi-Log Scale |

<sup>\*</sup> Depending on the number of subjects included in the PK population, the figure numbering presented here may change in the report.

<sup>\*\*</sup> Similar figures will be presented for each subject who received study medication



Zhejiang Teruisi Pharmaceutical Inc.

## **Table 2-3 List of Data Listings Shells**

| Listing<br>Number | Title |
|---|---|
| | Documentation of Statistical Methods |
| 16.1.9-1 | ANOVA for Treatment Comparisons (A/B, A/C and B/C) – PK Population |
| 16.1.9-2 | Wilcoxon Rank Sum Test for $T_{max}$ for Treatment Comparisons (A/B, A/C and B/C) – PK Population |
| | Subject Characteristics Listings |
| 16.2.1-1 | Subjects Completion and Discontinuation Information |
| 16.2.2-1 | Protocol Deviations |
| 16.2.4-1 | Demographics |
| 16.2.4-2 | Medical History Findings at Screening |
| 16.2.4-3 | Prior and Concomitant Medications |
| 16.2.4-4 | Study Drug Administration |
| | PK Data Listings |
| 16.2.6-1 | Listing of Individual Actual Sampling Times and Pharmacokinetic Concentrations |
| 16.2.6-2 | Listing of Individual Pharmacokinetic Parameters |
| | Safety Data Listings |
| 16.2.7-1 | Treatment-Emergent Adverse Events |
| 16.2.7-2 | Serious Adverse Events |
| 16.2.8-1 | Clinical Laboratory – Biochemistry |
| 16.2.8-2 | Clinical Laboratory – Hematology |
| 16.2.8-3 | Clinical Laboratory – Urinalysis |
| 16.2.8-4 | Vital Signs Result |
| 16.2.8-5 | Electrocardiogram Result |
| 16.2.8-6 | Immunogenicity Assessment |

Zhejiang Teruisi Pharmaceutical Inc.

## 3. CSR In-text Tables



**Table 10.1-1 Subject Disposition** 

| Category | TRS003, 3 mg/kg IV<br>Infusion Dose<br>(A) | China-Approved Bevacizumab,<br>3 mg/kg IV Infusion Dose<br>(B) | US Licensed Avastin <sup>®</sup> (Bevacizumab), 3 mg/kg IV Infusion Dose (C) | Overall |
|---|---|---|---|---|
| Screened | | | | XX |
| | - | - | - | |
| Screening Failures <sup>1,2</sup> | - | - | - | x ( xx.x) |
| Not Enrolled <sup>1,3</sup> | - | - | - | x ( xx.x) |
| Enrolled <sup>1,4</sup> | - | - | - | x ( xx.x) |
| Dosed | xx | XX | XX | XX |
| Not Dosed | xx | XX | XX | XX |
| Completed <sup>5</sup> | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| Number of Subjects Discontinued <sup>7</sup> Primary Reason for Discontinuation <sup>7, 8</sup> | xx | XX | XX | xx |
| Adverse Event | x ( xx.x) | x ( xx.x) | x ( xx.x) | x(xx.x) |
| Death | x ( xx.x) | x ( xx.x) | x ( xx.x) | x(xx.x) |
| Pregnancy | x ( xx.x) | x ( xx.x) | x ( xx.x) | x(xx.x) |
| Protocol Deviation | x ( xx.x) | x ( xx.x) | x ( xx.x) | x(xx.x) |
| Lost to Follow-up | x ( xx.x) | x ( xx.x) | x ( xx.x) | x(xx.x) |
| Study Terminated by Sponsor | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| Non-Compliance with Study Drug | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| Withdrawal by Subject | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| Physician Decision | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| Other | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |

 19-SEP-2018 (Final 1.0)

<sup>&</sup>lt;sup>1</sup> Percentage based on the number of screened subjects.
<sup>2</sup> Screening failures include volunteers who did not meet project criteria.

<sup>&</sup>lt;sup>3</sup> Not enrolled include volunteers who were judged eligible but decided not to participate on study or who were not selected to participate in the study since there was already a sufficient number of subjects.

<sup>&</sup>lt;sup>4</sup> Enrolled include volunteers who were judged eligible and accepted to participate in the trial after having signed the approved final version of the study informed consent



Zhejiang Teruisi Pharmaceutical Inc.

Data source: Listings 16.2.1-1 and 16.2.4-4.

19-SEP-2018 (Final 1.0) 

form and also those identified as standby who may replace subjects who withdraw from the study before dosing.

<sup>5</sup> Percentage based on the number of dosed subjects for a given treatment.

<sup>6</sup> Percentage based on the overall number of subjects dosed (safety population).

<sup>7</sup> Overall, each subject could only contribute once to each reason for discontinuation, regardless of the number of occurrences.

<sup>&</sup>lt;sup>8</sup> Percentage based on the number of discontinued subjects per treatment group or overall, as appropriate.



Zhejiang Teruisi Pharmaceutical Inc.

Table 11.4.2.3-1 Summary of Pharmacokinetic Parameters – PK Population

| Parameter (unit) | TRS003, 3 mg/kg IV Infusion Dose (A) | | | China-Approved Bevacizumab, 3 mg/kg IV<br>Infusion Dose<br>(B) | | | US Licensed Avastin <sup>®</sup> (Bevacizumab), 3 mg/kg IV Infusion Dose (C) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | Mean | SD | CV% | N Mean SD CV% | | | N Mean SD CV% | | | | |
| $\begin{array}{c} AUC_{0\text{-t}}\left(h^*pg/mL\right)\\ AUC_{0\text{-inf}}\left(h^*pg/mL\right)\\ Residual\ area\ (\%)\\ C_{max}\left(pg/mL\right)\\ T_{\frac{1}{2}\text{ el}}\left(h\right)\\ K_{\text{el}}\left(/h\right)\\ Cl\left(L/h\right)\\ V_{\text{d}}\left(L\right) \end{array}$ | | | | | | | | | | | | |
| | TH | RS003, 3 mg | | ıfusion | rsion China-Approved Bevacizuma Infusion Dose | | | 3 mg/kg IV | /kg IV US Licensed Avastin® (Bevacizumab). IV Infusion Dose | | | ab), 3 mg/kg |
| Parameter (unit) | | | Oose<br>(A) | | | | on Dose<br>(B) | | | | (C) | |
| i arameter (unit) | N | Median | Min | Max | N | Median | Min | Max | N | Median | Min | Max |
| T <sub>max</sub> (h) | | | | | | | | | | | | |

N: Number of observations; SD: Standard Deviation; CV%: Coefficient of Variation; Min: Minimum; Max: Maximum; '-': Not calculated.

19-SEP-2018 (Final 1.0) 



Zhejiang Teruisi Pharmaceutical Inc.

Table 11.4.2.3-2 Ratios (A/B and C/B), 90% Geometric Confidence Intervals, Inter-Subjects CV (%) and p-value – PK Population

| $ \begin{array}{c ccccccccccccccccccccccccccccccccccc$ | p-value | Inton Cubicat | eometric C.I. <sup>2</sup> | 90% G | Ratio <sup>1</sup> | ric LSM | Geomet | | Comparison |
|---|---|---|---|---|---|---|---|---|---|
| (h*pg/mL) $AUC_{0-inf}$ | Treatment | | | | | Trt2 | Trt1 | Parameter (unit) | (Trt1 vs Trt2) |
| | | | . , | | | | | | A vs B |
| $C_{max}$ (pg/mL) | | | | | | | | $C_{max} (pg/mL)$ | |

LSM: Least Square Mean; Trt: Treatment.

Probability (p) values are derived from Type III sums of squares; p-value for the treatment effect is tested against the residual mean square error.

Treatment A: TRS003, 3 mg/kg IV Infusion Dose; Treatment B: China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose;

Treatment C: US Licensed Avastin® (Bevacizumab), 3 mg/kg IV Infusion Dose.

Note: This table will be repeated for Table 11.4.2.3-3. Please adapt title and treatment footnotes accordingly.

19-SEP-2018 (Final 1.0) 

Calculated using least-squares means according to the formula:  $\exp^{(DIFFERENCE)} * 100$ .

2 90% Geometric Confidence Interval calculated according to the formula:  $\exp^{(DIFFERENCE \pm t)} * 100$ .

3 Calculated according to formula:  $\exp^{(MSE)} - 1$  \* 100.

Zhejiang Teruisi Pharmaceutical Inc.

## 4. Summary Tables



Table 14.1-1 Summary of Demographic Characteristics of Subjects Included in the Safety Population

| Category | Statistic | TRS003, 3 mg/kg IV Infusion<br>Dose<br>(A) | China-Approved Bevacizumab, 3 mg/kg IV<br>Infusion Dose<br>(B) | US Licensed Avastin® (Bevacizumab), 3 mg/kg IV Infusio Dose (C) |
|---|---|---|---|---|
| Age (years) | N | XX | XX | XX |
| | Mean | xx.x | XX.X | XX.X |
| | SD | xx.x | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX-XX | XX-XX | XX-XX |
| Age Groups | | | | |
| <18 | n (%) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| 18-40 | n (%) | x ( xx.x) | x ( xx.x) | x(xx.x) |
| > 40 | n (%) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| Ethnicity Not Hispanic or Latino | n (%) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| Hispanic or Latino | n (%) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| Race | | | | |
| White | n (%) | x ( xx.x) | x(xx.x) | x (xx.x) |
| Black | n (%) | x ( xx.x) | x(xx.x) | x ( xx.x) |
| Asian | n (%) | x ( xx.x) | x(xx.x) | x ( xx.x) |
| Am Indian | n (%) | x ( xx.x) | x(xx.x) | x ( xx.x) |
| Hawaiian | n (%) | x ( xx.x) | x(xx.x) | x (xx.x) |
| Multi-racial | n (%) | x ( xx.x) | x(xx.x) | x ( xx.x) |
| Other | n (%) | x ( xx.x) | x ( xx.x) | x(xx.x) |
| Height (cm) | N | XX | XX | XX |
| | Mean | xx.xx | xx.xx | xx.xx |
| | SD | XX.XX | xx.xx | XX.XX |
| | Median | XX.XX | xx.xx | XX.XX |
| | Min, Max | XX.XX-XX.XX | xx.xx-xx.xx | XX.XX-XX.XX |
| | · | | | |

19-SEP-2018 (Final 1.0) 



Zhejiang Teruisi Pharmaceutical Inc.

| Weight (kg) | N | XX | XX | XX |
|---|---|---|---|---|
| | Mean | xx.xx | xx.xx | XX.XX |
| | SD | XX.XX | xx.xx | XX.XX |
| | Median | xx.xx | xx.xx | XX.XX |
| | Min, Max | xx.xx-xx.xx | xx.xx-xx.xx | xx.xx-xx.xx |
| BMI (kg/m <sup>2</sup> ) | N | XX | XX | XX |
| | Mean | xx.xxx | XX.XXX | XX.XXX |
| | SD | XX.XXX | XX.XXX | XX.XXX |
| | Median | xx.xxx | XX.XXX | XX.XXX |
| | Min, Max | xx.xx-xx.xx | xx.xx-xx.xx | xx.xx-xx.xx |

## Programming Note:

1) Refer to the note below for additional instructions

N: Number of subjects dosed; n (%): Number and percent of subjects; SD: Standard Deviation.

Am Indian: American Indian or Alaskan Native; Black: Black or African American; Hawaiian: Native Hawaiian or Pacific Islander;

BMI: Body Mass Index.

Last results (scheduled or unscheduled) obtained at screening were used to generate this table.

Data source: Listing 16.2.4-1

Note: This table will be repeated for Table 14.1-2. Please adapt title and treatment footnotes accordingly.

19-SEP-2018 (Final 1.0) 



Zhejiang Teruisi Pharmaceutical Inc.

| Table 14.2.1-1 Descriptive Statistics for Bevacizumab | Plasma Concentration over N | Nominal Time by Treatme | ent – PK Population |
|---|---|---|---|
|---|---|---|---|

| Treatment | Nominal Time | Time Unit | N | Mean | SD | CV% | Min | Median | Max | Geometric Mean | Concentration Unit |
|---|---|---|---|---|---|---|---|---|---|---|---|
| A | Pre-dose | h | | | | | | | | | |
| | 0.000 (at EOI) | h | | | | | | | | | |
| | 0.500 | h | | | | | | | | | |
| | 4.00 | h | | | | | | | | | |
| | 8.00 | h | | | | | | | | | |
| | 24.0 | h | | | | | | | | | |
| | 48.0 | h | | | | | | | | | |
| | 96.0 | h | | | | | | | | | |
| | 168 | h | | | | | | | | | |
| | 336 | h | | | | | | | | | |
| | 672 | h | | | | | | | | | |
| | 1008 | h | | | | | | | | | |
| | 1344 | h | | | | | | | | | |
| | 1680 | h | | | | | | | | | |
| | 2016 | h | | | | | | | | | |

N: Number of observations; SD: Standard Deviation; CV%: Coefficient of Variation; Min: Minimum; Max: Maximum; '-': Not Calculated; EOI: End of infusion.

Treatment A: TRS003, 3 mg/kg IV Infusion Dose; Treatment B: China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose; Treatment C: US Licensed Avastin® (Bevacizumab), 3 mg/kg IV Infusion Dose.

Data source: Listing 16.2.6-1

19-SEP-2018 (Final 1.0) 



Zhejiang Teruisi Pharmaceutical Inc.

Table 14.2.1-2 Descriptive Statistics of Pharmacokinetic Parameters by Treatment – PK Population

| Treatment | Parameter(unit) | N | Mean | SD | CV% | Min | Median | Max | Geometric Mean |
|---|---|---|---|---|---|---|---|---|---|
| A | AUC <sub>0-t</sub> (pg*h/mL) | | | | | | | | |
| | $AUC_{0-inf}(pg*h/mL)$ | | | | | | | | |
| | Residual Area (%) | | | | | | | | |
| | $C_{max}$ (pg/mL) | | | | | | | | |
| | $T_{max}(h)$ | | | | | | | | |
| | $T_{1/2 el}(h)$ | | | | | | | | |
| | $K_{el}(/h)$ | | | | | | | | |
| | $K_{el Lower}(/h)$ | | | | | | | | |
| | $K_{el\ Upper}(/h)$ | | | | | | | | |
| | Cl (L/h) | | | | | | | | |
| | $V_{d}(L)$ | | | | | | | | |
| ••• | | | | | | | | | |

N: Number of observations; SD: Standard Deviation; CV%: Coefficient of Variation; Min: Minimum, Max: Maximum; '-': Not calculated.

Treatment A: TRS003, 3 mg/kg IV Infusion Dose; Treatment B: China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose;

Treatment C: US Licensed Avastin® (Bevacizumab), 3 mg/kg IV Infusion Dose.

Data source: Listing 16.2.6-2

19-SEP-2018 (Final 1.0) 



Zhejiang Teruisi Pharmaceutical Inc.

Table 14.2.1-3 Ratios (A/B, A/C and C/B), 90% Geometric Confidence Intervals, Inter-Subjects CV (%) and P-value – PK Population

| Commonicon | | Geomet | ric LSM | Ratio <sup>1</sup> | 90% Geo1 | metric C.I. <sup>2</sup> | Inter-Subject | p-value |
|---|---|---|---|---|---|---|---|---|
| Comparison<br>(Trt1 vs.Trt2) | Parameter(unit) | Trt1 | Trt2 | (Trt1/Trt2)<br>(%) | Lower (%) | Upper (%) | $CV (\%)^3$ | Treatment |
| A vs B | $\begin{aligned} &AUC_{0\text{-t}}\left(h^*pg/mL\right)\\ &AUC_{0\text{-inf}}\left(h^*pg/mL\right)\\ &C_{max}\left(pg/mL\right) \end{aligned}$ | | | | | | | |
| A vs C | $\begin{aligned} &AUC_{0t}\left(h*pg/mL\right)\\ &AUC_{0\inf}\left(h*pg/mL\right)\\ &C_{max}\left(pg/mL\right) \end{aligned}$ | | | | | | | |
| C vs B | $\begin{aligned} &AUC_{0\text{-t}}\left(h^*pg/mL\right)\\ &AUC_{0\text{-inf}}\left(h^*pg/mL\right)\\ &C_{max}\left(pg/mL\right) \end{aligned}$ | | | PEN/EV | | | | |

LSM: Least Square Mean; Trt: Treatment.

Treatment A: TRS003, 3 mg/kg IV Infusion Dose; Treatment B: China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose;

Treatment C: US Licensed Avastin<sup>®</sup> (Bevacizumab), 3 mg/kg IV Infusion Dose.

Data Source: Listing 16.1.9-1

19-SEP-2018 (Final 1.0) 

<sup>&</sup>lt;sup>1</sup>Calculated using least-squares means according to the formula: exp<sup>(DIFFERENCE)</sup> \* 100.

<sup>2</sup> 90% Geometric Confidence Interval calculated according to the formula: exp<sup>(DIFFERENCE ± t</sup> (dfResidual) \* SE DIFFERENCE) \* 100.

<sup>3</sup> Calculated according to formula: SQRT (exp (MSE) - 1) \* 100.



Table 14.3.1-1 Frequency of Subjects Experiencing Treatment-Emergent Adverse Events and Number of Events Summarized per Treatment – Safety Population

| MedDRA <sup>®</sup> System Organ Class<br>MedDRA <sup>®</sup> Preferred Term | Statistic | TRS003, 3 mg/kg IV Infusion Dose (N=XX) | China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose (N=XX) | US Licensed Avastin® (Bevacizumab),<br>3 mg/kg IV Infusion Dose<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|---|
| Number of TEAEs | E | XX | XX | XX | XX |
| Number of Subjects with TEAEs | n (%) | x ( xx.x) | x ( xx.x) | x (xx.x) | x (xx.x) |
| MedDRA <sup>®</sup> System Organ Class 1<br>MedDRA <sup>®</sup> Preferred Term 1<br>MedDRA <sup>®</sup> Preferred Term 2 | n(%) E<br>n(%) E<br>n(%) E | x ( xx.x) x<br>x ( xx.x) x<br>x ( xx.x) x | x ( xx.x) x<br>x ( xx.x) x<br>x ( xx.x) x | x ( xx.x) x<br>x ( xx.x) x<br>x ( xx.x) x | x ( xx.x) x<br>x ( xx.x) x<br>x ( xx.x) x |
| MedDRA® System Organ Class 2 | n(%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| MedDRA® Preferred Term 1<br>MedDRA® Preferred Term 2 | n(%) E<br>n(%) E | x ( xx.x) x<br>x ( xx.x) x | x ( xx.x) x<br>x ( xx.x) x | x ( xx.x) x<br>x ( xx.x) x | x ( xx.x) x<br>x ( xx.x) x |
| MedDRA® System Organ Class 3<br>MedDRA® Preferred Term 1<br>MedDRA® Preferred Term 2 | n(%) E<br>n(%) E<br>n(%) E | x ( xx.x) x<br>x ( xx.x) x<br>x ( xx.x) x | x ( xx.x) x<br>x ( xx.x) x<br>x ( xx.x) x | x ( xx.x) x<br>x ( xx.x) x<br>x ( xx.x) x | x ( xx.x) x<br>x ( xx.x) x<br>x ( xx.x) x |

## Programming Notes:

1) SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.

E: Number of TEAEs; N: Number of subjects dosed; n (%): Number and percent of subjects with TEAE; MedDRA®: Medical Dictionary for Regulatory Activities, version 21.0; TEAEs: Treatment-Emergent Adverse Events.

Each subject could only contribute once to each of the incidence rates, regardless of the number of occurrences.

Overall: Included results from all treatment groups.

Data source: Listing 16.2.7-1

19-SEP-2018 (Final 1.0) 

<sup>2)</sup> Refer to footnotes for additional instructions.



Zhejiang Teruisi Pharmaceutical Inc.

Table 14.3.1-2 Frequency of Subjects Experiencing Treatment-Emergent Adverse Events Summarized per Treatment and Severity – Safety Population

| MedDRA® System Organ Class | | | TRS003, 3 | mg/kg IV In | fusion Dose | | China-App | roved Beva | cizumab, 3 n | ng/kg IV Infi | usion Dose |
|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA® Preferred Term | | | | (N=XX) | | | | | (N=XX) | | |
| | n (%) | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| MedDRA® System Organ Class 1<br>MedDRA® Preferred Term 1<br>MedDRA® Preferred Term 2 | | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) |
| MedDRA <sup>®</sup> System Organ Class 2<br>MedDRA <sup>®</sup> Preferred Term 1<br>MedDRA <sup>®</sup> Preferred Term 2 | | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) |

#### Programming Notes:

- 1) SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.
- 2) If the distribution of treatments is presented on more than one page, preserve the order of the SOC and PT as defined in the generation of the global table without severity.
- 3) Refer to footnotes for additional instructions.

N: Number of subjects dosed; n (%): Number and percent of subjects with treatment-emergent adverse events; MedDRA®: Medical Dictionary for Regulatory Activities, version 21.0.

Each subject could only contribute once to each of the incidence rates, regardless of the number of occurrence; the highest severity is presented.

Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated; Grade 2: Moderate; minimal, local or non-invasive intervention indicated; limiting age-appropriate instrumental activities of daily; Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living; Grade 4: Life-threatening consequences; urgent intervention indicated; Grade 5: Death related to AE.

Overall: Included results from all treatment groups.

Data source: Listing 16.2.7-1

19-SEP-2018 (Final 1.0) 



Zhejiang Teruisi Pharmaceutical Inc.

Table 14.3.1-2 Frequency of Subjects Experiencing Treatment-Emergent Adverse Events Summarized per Treatment and Severity – Safety Population

| MedDRA® System Organ Class<br>MedDRA® Preferred Term | US License | US Licensed Avastin® (Bevacizumab), 3 mg/kg IV Infusion Dose $(N\!\!=\!\!XX)$ | | | | | | Overall (N=XX) | | |
|---|---|---|---|---|---|---|---|---|---|---|
| n (% | ) Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| MedDRA® System Organ Class 1 MedDRA® Preferred Term 1 MedDRA® Preferred Term 2 | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| MedDRA <sup>®</sup> System Organ Class 2 | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| MedDRA <sup>®</sup> Preferred Term 1 | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| MedDRA <sup>®</sup> Preferred Term 2 | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |

### Programming Notes:

- 1) SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.
- 2) If the distribution of treatments is presented on more than one page, preserve the order of the SOC and PT as defined in the generation of the global table without severity.
- 3) Refer to footnotes for additional instructions.

N: Number of subjects dosed; n (%): Number and percent of subjects with treatment-emergent adverse events; MedDRA®: Medical Dictionary for Regulatory Activities, version 21.0.

Each subject could only contribute once to each of the incidence rates, regardless of the number of occurrence; the highest severity is presented.

Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated; Grade 2: Moderate; minimal, local or non-invasive intervention indicated; limiting age-appropriate instrumental activities of daily; Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living; Grade 4: Life-threatening consequences; urgent intervention indicated; Grade 5: Death related to AE.

Overall: Included results from all treatment groups.

Data source: Listing 16.2.7-1

19-SEP-2018 (Final 1.0) 



Zhejiang Teruisi Pharmaceutical Inc.

Table 14.3.1-3 Number of Treatment-Emergent Adverse Events Summarized per Treatment and Severity – Safety Population

| MedDRA® System Organ Class | | | TRS003, 3 1 | mg/kg IV In | fusion Dose | | China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA® Preferred Term | | | (N=XX) | | | | (N=XX) | | | | |
| | Е | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| MedDRA® System Organ Class 1 | | X | X | X | X | X | X | X | X | X | X |
| MedDRA® Preferred Term 1 | | X | X | X | X | X | X | X | X | X | X |
| MedDRA® Preferred Term 2 | | X | X | X | X | X | X | X | X | X | X |
| MedDRA® System Organ Class 2 | | X | X | X | X | X | x | X | X | X | X |
| MedDRA® Preferred Term 1 | | X | X | X | X | X | x | X | x | X | X |
| MedDRA® Preferred Term 2 | | X | X | X | X | X | X | X | X | X | X |

### Programming Notes:

E: Number of treatment-emergent adverse event; N: Number of subjects dosed; MedDRA®: Medical Dictionary for Regulatory Activities, version 21.0.

Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated; Grade 2: Moderate; minimal, local or non-invasive intervention indicated; limiting age-appropriate instrumental activities of daily; Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living; Grade 4: Life-threatening consequences; urgent intervention indicated; Grade 5: Death related to AE.

Overall: Included results from all treatment groups.

Data source: Listing 16.2.7-1

19-SEP-2018 (Final 1.0) 

<sup>1)</sup> SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.

<sup>2)</sup> If the distribution of treatments is presented on more than one page, preserve the order of the SOC and PT as defined in the generation of the global table without severity.



Zhejiang Teruisi Pharmaceutical Inc.

Table 14.3.1-3 Number of Treatment-Emergent Adverse Events Summarized per Treatment and Severity – Safety Population

| MedDRA® System Organ Class<br>MedDRA® Preferred Term | | US Licensed | Avastin® (Be | evacizumab),<br>(N=XX) | 3 mg/kg IV I | nfusion Dose | Overall (N=XX) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Е | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| MedDRA <sup>®</sup> System Organ Class 1 | | x | x | x | x | x | X | X | X | x | x |
| MedDRA <sup>®</sup> Preferred Term 1 | | x | x | x | x | x | X | X | X | x | x |
| MedDRA <sup>®</sup> Preferred Term 2 | | x | x | x | x | x | X | X | X | x | x |
| MedDRA <sup>®</sup> System Organ Class 2 | | x | x | x | x | x | X | x | x | x | x |
| MedDRA <sup>®</sup> Preferred Term 1 | | x | x | x | x | x | X | x | x | x | x |
| MedDRA <sup>®</sup> Preferred Term 2 | | x | x | x | x | x | X | x | x | x | x |

### Programming Notes:

E: Number of treatment-emergent adverse event; N: Number of subjects dosed; MedDRA®: Medical Dictionary for Regulatory Activities, version 21.0.

Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated; Grade 2: Moderate; minimal, local or non-invasive intervention indicated; limiting age-appropriate instrumental activities of daily; Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living; Grade 4: Life-threatening consequences; urgent intervention indicated; Grade 5: Death related to AE.

Overall: Included results from all treatment groups.

Data source: Listing 16.2.7-1

19-SEP-2018 (Final 1.0) 

<sup>1)</sup> SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.

<sup>2)</sup> If the distribution of treatments is presented on more than one page, preserve the order of the SOC and PT as defined in the generation of the global table without severity.



Zhejiang Teruisi Pharmaceutical Inc.

Table 14.3.1-4 Frequency of Subjects Experiencing Treatment-Emergent Adverse Events Summarized per Treatment and Relationship – Safety Population

| MedDRA <sup>®</sup> System Organ Class<br>MedDRA <sup>®</sup> Preferred Term | TRS003, 3 mg/kg IV Infusion Dose (N=XX) | | Dose Bevacizumao, 3 mg/kg IV | | US Licensed Avastin <sup>®</sup> (Bevacizumab), 3 mg/kg IV Infusion Dose (N=XX) | | Overall (N=XX) | |
|---|---|---|---|---|---|---|---|---|
| n (%) | Related | Not Related | Related | Not Related | Related | Not Related | Related | Not Related |
| MedDRA® System Organ Class 1 | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| MedDRA® Preferred Term 1 | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| MedDRA® Preferred Term 2 | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| MedDRA® System Organ Class 2 | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| MedDRA® Preferred Term 1 | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| MedDRA® Preferred Term 2 | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |

#### Programming Notes:

N: Number of subjects dosed; n (%): Number and percent of subjects with treatment-emergent adverse event; MedDRA®: Medical Dictionary for Regulatory Activities, version 21.0.

Each subject could only contribute once to each of the incidence rates, regardless of the number of occurrence; the highest relationship is presented.

Overall: Included results from all treatment groups.

Data source: Listing 16.2.7-1

19-SEP-2018 (Final 1.0) 

<sup>1)</sup> SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.

<sup>2)</sup> If the distribution of treatments is presented on more than one page, preserve the order of the SOC and PT as defined in the generation of the global table without relationship.

<sup>3)</sup> Refer to footnotes for additional instructions.



Zhejiang Teruisi Pharmaceutical Inc.

Table 14.3.1-5 Number of Treatment-Emergent Adverse Events Summarized per Treatment and Relationship – Safety Population

| MedDRA® System Organ Class<br>MedDRA® Preferred Term | TRS003, 3 mg/kg IV Infusion Dose (N=XX) | | China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose (N=XX) | | US Licensed Avastin® (Bevacizumab), 3 mg/kg IV Infusion Dose (N=XX) | | Overall (N=XX) | |
|---|---|---|---|---|---|---|---|---|
| E | Related | Not Related | Related | Not Related | Related | Not Related | Related | Not Related |
| MedDRA® System Organ Class 1 | x | x | x | x | x | x | x | x |
| MedDRA® Preferred Term 1 | x | x | x | x | x | x | x | x |
| MedDRA® Preferred Term 2 | x | x | x | x | x | x | x | x |
| MedDRA® System Organ Class 2 | x | x | x | x | X | x | x | x |
| MedDRA® Preferred Term 1 | x | x | x | x | X | x | x | x |
| MedDRA® Preferred Term 2 | x | x | x | x | X | x | x | x |

#### Programming Notes:

E: Number of treatment-emergent adverse event; N: Number of subjects dosed; MedDRA®: Medical Dictionary for Regulatory Activities, version 21.0. Overall: Included results from all treatment groups.

Data source: Listing 16.2.7-1

19-SEP-2018 (Final 1.0) 

<sup>1)</sup> SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.

<sup>2)</sup> If the distribution of treatments is presented on more than one page, preserve the order of the SOC and PT as defined in the generation of the global table without relationship.



Zhejiang Teruisi Pharmaceutical Inc.

**Table 14.3.4-1 Biochemistry Summary Descriptive Statistics – Safety Population** 

| | | | | China-Approved Bevacizumab, 3 mg/kg | US Licensed Avastin® (Bevacizumab), 3 |
|---|---|---|---|---|---|
| Parameter (unit) | | | Dose | IV Infusion Dose | mg/kg IV Infusion Dose |
| Normal Range | Visit | Statistic | (N=XX) | (N=XX) | (N=XX) |
| Parameter 1 (unit) | Screening | n | XX | XX | XX |
| XX-XX | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | xx-xx | xx-xx |
| | Day -1 | n | XX | XX | xx |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | xx-xx | xx-xx |
| | Baseline | n | XX | XX | xx |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | xx-xx | xx-xx |
| | Day 2 | n | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | xx-xx | XX-XX |
| | Day 2 - CFB | n | XX | XX | xx |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | xx-xx | xx-xx |
| | Day 8 | n | XX | XX | xx |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | xx-xx | XX-XX | XX-XX |

19-SEP-2018 (Final 1.0) 



Zhejiang Teruisi Pharmaceutical Inc.

**Table 14.3.4-1 Biochemistry Summary Descriptive Statistics – Safety Population** 

| | | | | China-Approved Bevacizumab, 3 mg/kg | US Licensed Avastin® (Bevacizumab), |
|---|---|---|---|---|---|
| Parameter (unit) | | | Dose | IV Infusion Dose | mg/kg IV Infusion Dose |
| Normal Range | Visit | Statistic | (N=XX) | (N=XX) | (N=XX) |
| | Day 8 - CFB | n | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | XX-XX | xx-xx |
| | Day 29 | n | XX | XX | xx |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | xx.x | XX.X | XX.X |
| | | Median | xx.x | XX.X | XX.X |
| | | Min, Max | XX-XX | XX-XX | xx-xx |
| | Day 29 - CFB | n | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | XX-XX | xx-xx |
| | Day 57 | n | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | XX-XX | xx-xx |
| | Day 57 - CFB | n | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | xx-xx | xx-xx |
| | Day 85 (EOS) | n | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | xx-xx | XX-XX | XX-XX |

19-SEP-2018 (Final 1.0) 



Zhejiang Teruisi Pharmaceutical Inc.

**Table 14.3.4-1 Biochemistry Summary Descriptive Statistics – Safety Population** 

| Damamatan (unit) | | | TRS003, 3 mg/kg IV Infusion<br>Dose | China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose | US Licensed Avastin® (Bevacizumab), 3<br>mg/kg IV Infusion Dose |
|---|---|---|---|---|---|
| Parameter (unit) | | | | | 5 5 |
| Normal Range | Visit | Statistic | (N=XX) | (N=XX) | (N=XX) |
| | Day 85 (EOS) - CFB | n | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | XX-XX | XX-XX |

CFB: Change from baseline; N: Number of subjects dosed; n: Number of subjects; SD: Standard Deviation; EOS: End of study.

Baseline is defined as the last results (scheduled or unscheduled) obtained prior to infusion.

Data source: Listing 16.2.8-1

Note: This table will be repeated for Tables 14.3.4-3, and 14.3.4-5. Please adapt title and footnotes accordingly.

19-SEP-2018 (Final 1.0) 



Zhejiang Teruisi Pharmaceutical Inc.

Table 14.3.4-2 Frequency of Subjects – Biochemistry Shifts from Baseline – Safety Population

| | Baseline Flag: | | Low | | | Normal | | | High | |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Post-Baseline Flag: | Low | Normal | High | Low | Normal | High | Low | Normal | High |
| Parameter (unit) | Visit | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| TRS003, 3 mg/kg IV Infusion Dose | | | | | | | | | | |
| (N=XX) | | | | | | | | | | |
| Parameter 1 | Day 2 | x (xx.x) | x(xx.x) | x(xx.x) | x (xx.x) | x(xx.x) | x(xx.x) | x (xx.x) | x (xx.x) | x(xx.x) |
| | Day 8 | x (xx.x) | x(xx.x) | x(xx.x) | x (xx.x) | x(xx.x) | x(xx.x) | x (xx.x) | x(xx.x) | x(xx.x) |
| | Day 29 | x (xx.x) | x(xx.x) | x(xx.x) | x (xx.x) | x(xx.x) | x(xx.x) | x (xx.x) | x(xx.x) | x(xx.x) |
| | Day 57 | x (xx.x) | x(xx.x) | x(xx.x) | x (xx.x) | x(xx.x) | x(xx.x) | x (xx.x) | x(xx.x) | x(xx.x) |
| | Day 85 (EOS) | x (xx.x) | x(xx.x) | x(xx.x) | x (xx.x) | x(xx.x) | x(xx.x) | x (xx.x) | x (xx.x) | x ( xx.x) |
| Parameter 2 | Day 2<br>Day 8<br>Day 29<br>Day 57<br>Day 85 (EOS) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x (xx.x)<br>x (xx.x)<br>x (xx.x)<br>x (xx.x)<br>x (xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) |
| <br>Add for all other Treatments and<br>Parameters | | | | | | | | | | |

### Programming Notes:

- 1) Preserve parameters, scheduled visits and sorting defined in Summary Descriptive Statistics Table
- 2) Refer to footnotes for additional instructions.
- 3) Adapt Data Source to the appropriate laboratory category listing.

N: Number of subjects dosed; n: Number and percent of subjects; EOS: End of study.

Baseline is defined as the last results (scheduled or unscheduled) obtained prior to infusion.

Percentage based on the number of subjects having available results at baseline and at the specific post-baseline visit.

Data source: Listing 16.2.8-1

Note: This table will be repeated for Tables 14.3.4-4, and 14.3.4-6. Please adapt title and footnotes accordingly.

19-SEP-2018 (Final 1.0) 



Zhejiang Teruisi Pharmaceutical Inc.

| Parameter (unit)<br>Normal Range | Visit | Result n (%) | TRS003, 3 mg/kg IV Infusion<br>Dose<br>(N=XX) | China-Approved Bevacizumab, 3<br>mg/kg IV Infusion Dose<br>(N=XX) | US Licensed Avastin®<br>(Bevacizumab), 3 mg/kg IV<br>Infusion Dose<br>(N=XX) |
|---|---|---|---|---|---|
| Parameter 1(unit) | Screening | Negative | x (xx.x) | x(xx.x) | x (xx.x) |
| XX-XX | | Trace | x (xx.x) | x (xx.x) | x(xx.x) |
| | Day -1 | Negative | x (xx.x) | x (xx.x) | x (xx.x) |
| | | Trace | x (xx.x) | x (xx.x) | x (xx.x) |
| | Baseline | Negative | x (xx.x) | x (xx.x) | x (xx.x) |
| | | Trace | x(xx.x) | x (xx.x) | x (xx.x) |
| | Day 2 | Negative | x (xx.x) | x (xx.x) | x (xx.x) |
| | • | Trace | x(xx.x) | x (xx.x) | x (xx.x) |
| | Day 8 | Negative | x (xx.x) | x (xx.x) | x (xx.x) |
| | · | Trace | x(xx.x) | x (xx.x) | x (xx.x) |
| | Day 29 | Negative | x (xx.x) | x (xx.x) | x (xx.x) |
| | • | Trace | x (xx.x) | x (xx.x) | x (xx.x) |
| | Day 57 | Negative | x (xx.x) | x (xx.x) | x (xx.x) |
| | - | Trace | x (xx.x) | x(xx.x) | x (xx.x) |
| | Day 85 (EOS) | Negative | x (xx.x) | x (xx.x) | x (xx.x) |
| | <b>3</b> - ( ) | Trace | x (xx.x) | x(xx.x) | x(xx.x) |

#### Programming Notes:

- 1) Urine Microscopy parameters will not presented in this table.
- 2) Evaluate if the units must be added to parameter name if a numeric result was observed. Remove (units) from column header if no numeric results were observed.
- 3) For each parameter provide normal range of primary facility and, for gender specific parameters, use the same sorting of gender from demographic table.
- 4) Independently for each parameter, sort results by gradation.
- 5) Refer to footnotes for additional instructions.

N: Number of subjects dosed; n (%): Number and percent of subjects; EOS: End of study.

Percentage based on the number of subjects having available result at each visit, independently for each parameter.

Data source: Listing 16.2.8-3



Table 14.3.4-8 Frequency of Subjects – Urinalysis Shifts from Screening – Categorical Results – Safety Population

| | Baseline Flag: | Nor | mal | Abnormal | |
|---|---|---|---|---|---|
| Treatment | Post-Baseline Flag: | Normal | Abnormal | Normal | Abnormal |
| Parameter (unit) | Visit | n (%) | n (%) | n (%) | n (%) |
| TRS003, 3 mg/kg IV Infusion Dose (N=XX) | | | | | |
| Parameter 1 | Day 2 | x(xx.x) | x (xx.x) | x(xx.x) | x(xx.x) |
| | Day 8 | x(xx.x) | x (xx.x) | x(xx.x) | x(xx.x) |
| | Day 29 | x(xx.x) | x (xx.x) | x(xx.x) | x(xx.x) |
| | Day 57 | x(xx.x) | x(xx.x) | x(xx.x) | x(xx.x) |
| | Day 85 (EOS) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| Parameter 2 | Day 2 | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| | Day 8 | x(xx.x) | x (xx.x) | x(xx.x) | x(xx.x) |
| | Day 29 | x(xx.x) | x (xx.x) | x(xx.x) | x(xx.x) |
| | Day 57 | x(xx.x) | x (xx.x) | x(xx.x) | x(xx.x) |
| | Day 85 (EOS) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| Add for all other Treatments and Parameters | | | | | |

#### Programming Notes:

- 1) Preserve parameters, scheduled visits and sorting defined in Summary Descriptive Statistics Table
- 2) Refer to footnotes for additional instructions.
- 3) Adapt Data Source to the appropriate laboratory category listing.

N: Number of subjects dosed; n: Number and percent of subjects; EOS: End of study.

Baseline is defined as the last results (scheduled or unscheduled) obtained prior to Infusion.

Percentage based on the number of subjects having available results at baseline and at the specific post-baseline visit.

Data source: Listing 16.2.8-3

19-SEP-2018 (Final 1.0) 



Zhejiang Teruisi Pharmaceutical Inc.

**Table 14.3.4-9 Vital Signs Summary Descriptive Statistics – Safety Population** 

| | | | | China-Approved Bevacizumab, 3 mg/kg | US Licensed Avastin® (Bevacizumab), |
|---|---|---|---|---|---|
| Parameter (unit) | | | Dose | IV Infusion Dose | mg/kg IV Infusion Dose |
| Normal Range | Timepoint | Statistic | (N=XX) | (N=XX) | (N=XX) |
| Parameter 1 (unit) | Screening | n | XX | XX | XX |
| XX-XX | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | xx-xx | xx-xx |
| | Day -1 | n | XX | XX | xx |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | xx-xx | xx-xx |
| | Day 1, Pre-dose | n | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | xx-xx | xx-xx |
| | Baseline | n | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | xx-xx | xx-xx |
| | 0H Infusion | n | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | xx-xx | xx-xx |
| | 0H Infusion - CFB | n | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | xx-xx | XX-XX | XX-XX |

19-SEP-2018 (Final 1.0) 



Zhejiang Teruisi Pharmaceutical Inc.

**Table 14.3.4-9 Vital Signs Summary Descriptive Statistics – Safety Population** 

| Parameter (unit) | | | TRS003, 3 mg/kg IV Infusion Dose | China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose | US Licensed Avastin® (Bevacizumab), mg/kg IV Infusion Dose |
|---|---|---|---|---|---|
| Normal Range | Timepoint | Statistic | (N=XX) | (N=XX) | (N=XX) |
| | 0H (Post EOI) | n | xx | XX | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | xx-xx | XX-XX |
| | 0H (Post EOI) - CFB | n | XX | xx | XX |
| | · | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | xx-xx | xx-xx |
| | 0.5H (Post EOI) | n | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | xx-xx | xx-xx |
| | 0.5H (Post EOI) - CFB | n | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | xx-xx | xx-xx |
| | 4H, Day 1 | n | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | XX-XX | XX-XX |
| | 4H, Day 1 - CFB | n | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | XX-XX | XX-XX |

19-SEP-2018 (Final 1.0) 



Zhejiang Teruisi Pharmaceutical Inc.

**Table 14.3.4-9 Vital Signs Summary Descriptive Statistics – Safety Population** 

| | | | | China-Approved Bevacizumab, 3 mg/kg | US Licensed Avastin® (Bevacizumab), 3 |
|---|---|---|---|---|---|
| Parameter (unit) | | | Dose | IV Infusion Dose | mg/kg IV Infusion Dose |
| Normal Range | Timepoint | Statistic | (N=XX) | (N=XX) | (N=XX) |
| | 8H, Day 1 | n | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | xx-xx | xx-xx |
| | 8H Day 1 - CFB | n | XX | XX | XX |
| | - | Mean | XX.X | XX.X | XX.X |
| | | SD | xx.x | XX.X | XX.X |
| | | Median | xx.x | XX.X | XX.X |
| | | Min, Max | XX-XX | XX-XX | XX-XX |
| | Day 2 | n | xx | XX | XX |
| Day 2 | Duy 2 | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X<br>XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | XX-XX | XX-XX |
| | Day 2 - CFB | n | XX | xx | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | xx-xx | xx-xx |
| | Day 3 | n | XX | XX | xx |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | xx-xx | xx-xx |
| | Day 3 - CFB | n | XX | xx | xx |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | XX-XX | XX-XX |

19-SEP-2018 (Final 1.0) 



Zhejiang Teruisi Pharmaceutical Inc.

**Table 14.3.4-9 Vital Signs Summary Descriptive Statistics – Safety Population** 

| | | | | China-Approved Bevacizumab, 3 mg/kg | US Licensed Avastin® (Bevacizumab), |
|---|---|---|---|---|---|
| Parameter (unit) | | | Dose | IV Infusion Dose | mg/kg IV Infusion Dose |
| Normal Range | Timepoint | Statistic | (N=XX) | (N=XX) | (N=XX) |
| | <b>D</b> 0 | | | | |
| | Day 8 | n | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | XX-XX | XX-XX |
| | Day 8 - CFB | n | XX | XX | XX |
| | | Mean | xx.x | XX.X | XX.X |
| | | SD | xx.x | XX.X | XX.X |
| | | Median | xx.x | XX.X | XX.X |
| | | Min, Max | XX-XX | xx-xx | xx-xx |
| | Day 29 | n | XX | xx | xx |
| y | <b>y</b> - | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | xx-xx | xx-xx |
| | Day 29 - CFB | n | XX | xx | XX |
| | Duy 27 CI B | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X<br>XX.X | XX.X<br>XX.X | XX.X |
| | | Min, Max | XX-XX | XX-XX | XX-XX |
| | Day 57 | , | VV | XX | XX |
| | Day 37 | n<br>Mean | XX | | |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | XX-XX | XX-XX |
| | Day 57 - CFB | n | XX | XX | xx |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | xx-xx | XX-XX | XX-XX |

19-SEP-2018 (Final 1.0) 


Zhejiang Teruisi Pharmaceutical Inc.

Table 14.3.4-9 Vital Signs Summary Descriptive Statistics – Safety Population

| Parameter (unit) | | | TRS003, 3 mg/kg IV Infusion<br>Dose | China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose | US Licensed Avastin <sup>®</sup> (Bevacizumab), 3<br>mg/kg IV Infusion Dose |
|---|---|---|---|---|---|
| Normal Range | Timepoint | Statistic | (N=XX) | (N=XX) | (N=XX) |
| | Day 85 (EOS) | n | xx | xx | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | XX-XX | XX-XX |
| | Day 85 (EOS) - CFB | n | XX | XX | xx |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | XX-XX | XX-XX |

CFB: Change from baseline; N: Number of subjects dosed; n: Number of subjects; SD: Standard Deviation; EOS: End of study; EOI: End of infusion.

Baseline is defined as the last results (scheduled or unscheduled) obtained prior to infusion.

Data source: Listing 16.2.8-4

19-SEP-2018 (Final 1.0) 



Zhejiang Teruisi Pharmaceutical Inc.

Table 14.3.4-10 Electrocardiogram Summary Descriptive Statistics – Safety Population

| | | | TRS003, 3 mg/kg IV Infusion | China-Approved Bevacizumab, 3 mg/kg | US Licensed Avastin® (Bevacizumab), 3 |
|---|---|---|---|---|---|
| Parameter (unit) | | | Dose | IV Infusion Dose | mg/kg IV Infusion Dose |
| Normal Range | Timepoint | Statistic | (N=XX) | (N=XX) | (N=XX) |
| Parameter 1 (unit) | Screening | n | XX | XX | XX |
| XX-XX | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | xx-xx | xx-xx |
| | 0.5H (Post EOI) | n | XX | xx | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | xx-xx | xx-xx |
| | 0.5H (Post EOI) - CFS | n | XX | XX | xx |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | XX-XX | XX-XX |
| | Day 85 (EOS) | n | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX-XX | xx-xx | xx-xx |
| | Day 85 (EOS) - CFS | n | XX | xx | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | xx-xx | XX-XX | XX-XX |

CFS: Change from screening; N: Number of subjects dosed; n: Number of subjects; SD: Standard Deviation; EOS: End of study; EOI: End of infusion. Screening is defined as the last screened results (scheduled or unscheduled).

Data source: Listing 16.2.8-5

19-SEP-2018 (Final 1.0) 



Zhejiang Teruisi Pharmaceutical Inc.

**Table 14.3.4-11 Descriptive Statistics of Immunogenicity - Safety Population** 

| | | | | - F | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Nominal Time | Time Unit | N | Mean | SD | CV% | Min | Median | Max | Result Unit |
| 0.000 | h | | | | | | | | |
| 336 | h | | | | | | | | |
| 672 | h | | | | | | | | |
| 1344 | h | | | | | | | | |
| 2016 | h | | | | | | | | |
| | Nominal Time<br>0.000<br>336<br>672<br>1344 | Nominal Time Time Unit 0.000 h 336 h 672 h 1344 h | Nominal Time Time Unit N | Nominal Time Time Unit N Mean 0.000 h 336 h 672 h 1344 h | Nominal Time Time Unit N Mean SD 0.000 h 336 h 672 h 1344 h | Nominal Time Time Unit N Mean SD CV% 0.000 h 336 h 672 h 1344 h | Nominal Time Time Unit N Mean SD CV% Min 0.000 h 336 h 672 h 1344 h | Nominal Time Time Unit N Mean SD CV% Min Median 0.000 h 336 h 672 h 1344 h | 0.000 h 336 h 672 h 1344 h |

. . .

N: Number of observations; SD: Standard Deviation; CV%: Coefficient of Variation; Min: Minimum, Max: Maximum. Treatment A: TRS003, 3 mg/kg IV Infusion Dose; Treatment B: China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose;

Treatment C: US Licensed Avastin® (Bevacizumab), 3 mg/kg IV Infusion Dose.

Data source: Listing 16.2.8-6

19-SEP-2018 (Final 1.0) 

Zhejiang Teruisi Pharmaceutical Inc.

# 5. Figures



Figure 14.2.2-1a: Plasma Concentrations for Subject XX - Linear Scale



Treatment A: TRS003, 3 mg/kg IV Infusion Dose; Treatment B: China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose; Treatment C: US Licensed Avastin<sup>®</sup> (Bevacizumab), 3 mg/kg IV Infusion Dose.



Figure 14.2.2-1b: Plasma Concentrations for Subject XX – Semi-Log Scale



Treatment A: TRS003, 3 mg/kg IV Infusion Dose; Treatment B: China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose; Treatment C: US Licensed Avastin<sup>®</sup> (Bevacizumab), 3 mg/kg IV Infusion Dose.



Figure 14.2.2-115a: Mean (± SD) Plasma Concentrations - Linear Scale



Treatment A: TRS003, 3 mg/kg IV Infusion Dose; Treatment B: China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose; Treatment C: US Licensed Avastin® (Bevacizumab), 3 mg/kg IV Infusion Dose.



Figure 14.2.2-115b: Mean (± SD) Plasma Concentrations - Semi-Log Scale



Treatment A: TRS003, 3 mg/kg IV Infusion Dose; Treatment B: China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose; Treatment C: US Licensed Avastin<sup>®</sup> (Bevacizumab), 3 mg/kg IV Infusion Dose.



Figure 14.2.2-116a: Overlay of Individual and Mean Plasma Concentrations by Treatment - Linear Scale



Treatment A: TRS003, 3 mg/kg IV Infusion Dose; Treatment B: China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose; Treatment C: US Licensed Avastin<sup>®</sup> (Bevacizumab), 3 mg/kg IV Infusion Dose.



Figure 14.2.2-116b: Overlay of Individual and Mean Plasma Concentrations by Treatment - Semi-Log Scale



Treatment A: TRS003, 3 mg/kg IV Infusion Dose; Treatment B: China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose; Treatment C: US Licensed Avastin<sup>®</sup> (Bevacizumab), 3 mg/kg IV Infusion Dose.

Zhejiang Teruisi Pharmaceutical Inc.

# 6. Listings

Zhejiang Teruisi Pharmaceutical Inc.

# Listing 16.1.9-1 ANOVA for Treatment Comparisons (A/B, A/C and B/C) – PK Population

### The GLM Procedure

### Comparison: A vs B; Parameter: xxxx (unit).

| Class | Levels Values |
|-----------|----------------------|
| TRT | |
| Number o | of Observations Read |
| Number of | of Observations Used |

# The GLM Procedure Dependent Variable: LN\_AUCLST

| Source | DF | Sum of Squares | Mean S | quare I | F Value | Pr > F |
|---|---|---|---|---|---|---|
| Model | , | , | | | ٠ | |
| Error | | | | | | |
| Corrected Total | | | | | | |
| <del>-</del> | R-Square | Coeff Var | Root MSE | VAR Me | an | |
| Source | DF | Type III SS | Mean S | Square | F Value | Pr > I |
| TRT | | | | | | |
| | | The GLM Pr | ocedure | | | |
| Source | Type III Exp | pected Mean Squa | re | | | |
| ΓRT | Var(Error) | 2 Var(subject) | | | | |

### The GLM Procedure

## Tests of Hypotheses for Mixed Model Analysis of Variance Dependent Variable: LN\_AUCLST

| Source | DF Type III SS | Mean Square | F Value | Pr > F |
|--------|----------------|-------------|---------|--------|



Zhejiang Teruisi Pharmaceutical Inc.

| Source | | DF | Type III SS | S Mea | n Square | F Value | Pr > F |
|---|---|---|---|---|---|---|---|
| TRT | | | | | | | |
| Error: MS( | Error) | | | | | | |
| | | | Least S | Squares M | leans | | |
| | | | | | H0:LSM | ean1=LSMean2 | |
| TRTVAR | LSMEAN | | | | | | Pr > t |
| A | | | | | | | |
| В | | | | | | | |
| TRT VAR | LSMEAN | | | | 90% | Confidence Limits | |
| A | LSWILAN | | | | 7070 | Confidence Limits | |
| В | | | | | | | |
| Least Squa | res Means for | : Effec | t Treatment | | | | |
| i j Dit | fference Betw | een M | eans C | 00% Confide | ence Limits | for LSMean(i)-LSM | lean(i) |
| . , | reference Bern | CC11 1V1 | cuiis | o o o connac | nice Emme | Tor Estitedit(1) Estit | (Curity) |
| 1 2 | | | | | | | |
| | | D | | | A TIC | ICT | |
| | - | Depe | ndent Va | riable: Li | N_AUC | LSI | |
| | | St | andard | | | | |
| Parameter | Estimate | | rror | t Value | Pr > t | 90% Confidence L | imits |
| A-B | | | | | | | |

Treatment A: TRS003, 3 mg/kg IV Infusion Dose; Treatment B: China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose; Treatment C: US Licensed Avastin<sup>®</sup> (Bevacizumab), 3 mg/kg IV Infusion Dose.

Note: All ANOVA results for ln-transformed  $AUC_{0\text{-t}}$ ,  $AUC_{0\text{-inf}}$ , and  $C_{max}$  and untransformed  $T_{max}$ ,  $K_{el}$ , and  $T_{1/2\ el}$  will be presented for treatment A vs treatment C and treatment B vs treatment C comparisons in this listing.

Zhejiang Teruisi Pharmaceutical Inc.

Listing 16.1.9-2 Wilcoxon Rank Sum Test for  $T_{max}$  for Treatment Comparison (A/B, A/C and B/C) – PK Population

| and Brey Tix Topulation | | |
|-------------------------|-----------|-------|
| Difference | Statistic | Value |
| A - B | n | |
| | Mean | |
| | Median | |
| | SD | |
| | Min | |
| | Max | |
| Wilcoxon | S | |
| Rank-Sum Test | p-value | |

n: Number of subjects; SD: Standard Deviation; Min: Minimum; Max: Maximum.

Treatment A: TRS003, 3 mg/kg IV Infusion Dose; Treatment B: China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose; Treatment C: US Licensed Avastin® (Bevacizumab), 3 mg/kg IV Infusion Dose.

Note: Wilcoxon Rank sum test for  $T_{max}$  will be also presented for treatment A vs treatment C and treatment B vs treatment C comparisons in this listing.



Zhejiang Teruisi Pharmaceutical Inc.

| <b>Listing 16.2.1-1 Subjects Completion and Discontinuation Information</b> |
|-----------------------------------------------------------------------------|
|-----------------------------------------------------------------------------|

| Subject | Treatment | Completion/ Discontinuation Date and Time | Primary Reason for Discontinuation | Comment |
|---|---|---|---|---|
| 001 | A | DD-MM-YYYYTHH:MM | XXX | XXX |

Treatment A: TRS003, 3 mg/kg IV Infusion Dose; Treatment B: China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose; Treatment C: US Licensed Avastin<sup>®</sup> (Bevacizumab), 3 mg/kg IV Infusion Dose.



Zhejiang Teruisi Pharmaceutical Inc.

| Listing | 16.2.2-1 | <b>Protocol</b> | <b>Deviations</b> |
|---------|----------|-----------------|-------------------|
|---------|----------|-----------------|-------------------|

| Subject Treatment Category D | Deviation |
|------------------------------|-----------|
|------------------------------|-----------|

Treatment A: TRS003, 3 mg/kg IV Infusion Dose; Treatment B: China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose; Treatment C: US Licensed Avastin® (Bevacizumab), 3 mg/kg IV Infusion Dose.



Zhejiang Teruisi Pharmaceutical Inc.

**Listing 16.2.4-1 Demographics** 

| Subject | Treatment | Age (years) | Race | Ethnicity | BMI (kg/m <sup>2</sup> ) | Height (cm) | Weight (kg) |
|---|---|---|---|---|---|---|---|

001 Α

BMI: Body Mass Index.

Last results (scheduled or unscheduled) obtained at screening were used to generate this table.

Treatment A: TRS003, 3 mg/kg IV Infusion Dose; Treatment B: China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose; Treatment C: US Licensed Avastin® (Bevacizumab), 3 mg/kg IV Infusion Dose.

 19-SEP-2018 (Final 1.0)



Zhejiang Teruisi Pharmaceutical Inc.

## **Listing 16.2.4-2 Medical History Findings at Screening**

| Subject | Treatment | Finding | MedDRA® Preferred Term | MedDRA® System Organ Class | Onset Date | Resolution Date (or Ongoing) |
|---|---|---|---|---|---|---|
| | | FINDING 1 | Preferred Term 1 | SOC 1 | YYYY-MM-DDTHH:MM | YYYY-MM-DDTHH:MM |
| | | FINDING 2 | Preferred Term 2 | SOC 2 | YYYY-MM-DDTHH:MM | ONGOING |

#### Programming Notes:

- 1) SOC and Finding will be presented in uppercase. The Preferred Term will be presented in "propercase". The SAS coding "/~n" between terms will generate the break line.
- 2) The SAS coding "/~n" between dates will generate the break line.
- 3) If finding is ongoing, replace missing resolution date per ONGOING.
- 4) Sort events per Subject, Start Date, Stop Date, SOC and PT.
- 5) For incomplete date display, refer to CDISC SDTM Implementation Guide according to ISO 8601 format.

MedDRA®: Medical Dictionary for Regulatory Activities; MedDRA® Version 21.0.

Treatment A: TRS003, 3 mg/kg IV Infusion Dose; Treatment B: China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose;

Treatment C: US Licensed Avastin® (Bevacizumab), 3 mg/kg IV Infusion Dose.

19-SEP-2018 (Final 1.0) 



Zhejiang Teruisi Pharmaceutical Inc.

**Listing 16.2.4-3 Prior and Concomitant Medications** 

| Treatment | Prior/ | WHO DDE ATC /<br>WHO DDE Preferred Term / | Dose (unit)/ | | Onset Date and Time/<br>Resolution Date and Time | Indication |
|---|---|---|---|---|---|---|
| Subject | Concomitant | Medication | Frequency | Route | (or Ongoing) | (Condition or AE No.) |
| A | Prior | ATC 1/<br>Preferred Term 1/<br>MEDICATION 1/ | 20 (mg)<br>QID | ORAL | YYYY-MM-DDTHH:MM/<br>YYYY-MM-DDTHH:MM | |
| В | Concomitant | ATC 2/<br>Preferred Term 2/<br>MEDICATION 2/ | | | YYYY-MM-DDTHH:MM/<br>ONGOING | |

#### Programming Notes:

- 1) ATC and Medication will be presented in uppercase. The Preferred Term will be presented in "propase". The SAS coding "/~n" between terms will generate the break line.
- 2) The SAS coding "/~n" will generate the break line between treatment sequence and treatment, dose with units and frequency. In the same way apply a break line between dates.
- 3) If medication is ongoing, replace missing resolution date per ONGOING.
- 4) Sort events per Subject, Onset Date, Resolution Date, ATC and PT.
- 5) For incomplete date display, refer to CDISC SDTM Implementation Guide according to ISO 8601 format.

ATC: Anatomic Therapeutic Chemical; WHO DDE: World Health Organization Drug Dictionary Enhanced Version Mar2018, format B.

Treatment A: TRS003, 3 mg/kg IV Infusion Dose; Treatment B: China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose;

Treatment C: US Licensed Avastin<sup>®</sup> (Bevacizumab), 3 mg/kg IV Infusion Dose.

19-SEP-2018 (Final 1.0) 



Zhejiang Teruisi Pharmaceutical Inc.

## **Listing 16.2.4-4 Study Drug Administration**

| | ··-·· | | | |
|---|---|---|---|---|
| Subject | Treatment | Infusion Start Date and Time | Infusion End Date and Time | Total Dose |

YYYY-MM-DDTHH:MM:SS

Treatment A: TRS003, 3 mg/kg IV Infusion Dose; Treatment B: China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose; Treatment C: US Licensed Avastin<sup>®</sup> (Bevacizumab), 3 mg/kg IV Infusion Dose.

YYYY-MM-DDTHH:MM:SS

 19-SEP-2018 (Final 1.0)



Zhejiang Teruisi Pharmaceutical Inc.

Listing 16.2.6-1 Listing of Individual Actual Sampling Times and Pharmacokinetic Concentrations

| | | | concentration | Concentration Unit | Excluded Flag | Reason | Dose Date and Time | PK Sampling Date and Time |
|---|---|---|---|---|---|---|---|---|
| Pre-dose | h | 0.005 | | na/mI | N | | DDMMMYYYYT | DDMMMYYYYT |
| Pre-dose | h | 0.005 | | pg/mL | IN | | HH:MM:SS | HH:MM:SS |
| 0.000 (at EOI) | h | 0.001 | | pg/mL | N | | | |
| 0.500 | h | 0.489 | | pg/mL | Y | inconclusive | | |
| 4.00 | h | 4.001 | | | | | | |
| ••• | | | | | | | | |
| Pre-dose | h | 0.005 | | pg/mL | N | | | |
| 0.000 (at EOI) | h | 0.001 | | pg/mL | N | | | |
| 0.500 | h | 0.489 | | pg/mL | Y | inconclusive | | |
| 4.00 | h | 4.001 | | | | | | |
| | 0.500<br>4.00<br><br>Pre-dose<br>0.000 (at EOI)<br>0.500 | 4.00 h Pre-dose h 0.000 (at EOI) h 0.500 h | 0.500 h 0.489 4.00 h 4.001 Pre-dose h 0.005 0.000 (at EOI) h 0.001 0.500 h 0.489 | 0.500 h 0.489 4.00 h 4.001 Pre-dose h 0.005 0.000 (at EOI) h 0.001 0.500 h 0.489 | 0.500 h 0.489 pg/mL 4.00 h 4.001 Pre-dose h 0.005 pg/mL 0.000 (at EOI) h 0.001 pg/mL 0.500 h 0.489 pg/mL | 0.500 h 0.489 pg/mL Y 4.00 h 4.001 Pre-dose h 0.005 pg/mL N 0.000 (at EOI) h 0.001 pg/mL N 0.500 h 0.489 pg/mL Y | 0.500 h 0.489 pg/mL Y inconclusive 4.00 h 4.001 Pre-dose h 0.005 pg/mL N 0.000 (at EOI) h 0.001 pg/mL N 0.500 h 0.489 pg/mL Y inconclusive | 0.000 (at EOI) h 0.001 pg/mL N 0.500 h 0.489 pg/mL Y inconclusive 4.00 h 4.001 Pre-dose h 0.005 pg/mL N 0.000 (at EOI) h 0.001 pg/mL N 0.500 h 0.489 pg/mL Y inconclusive |

EOI: End of infusion.

Treatment A: TRS003, 3 mg/kg IV Infusion Dose; Treatment B: China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose; Treatment C: US Licensed Avastin® (Bevacizumab), 3 mg/kg IV Infusion Dose.

 19-SEP-2018 (Final 1.0)



Zhejiang Teruisi Pharmaceutical Inc.

Listing 16.2.6-2 Listing of Individual Pharmacokinetic Parameters

| Subject | Treatment | Parameter | Results | Unit | Excluded Flag | Reason |
|---|---|---|---|---|---|---|
| 001 | A | AUC <sub>0-t</sub> | | | N | |
| | | $\mathrm{AUC}_{0	ext{-inf}}$ | | | N | |
| | | $C_{max}$ | | | Y | Not Estimable |
| | | Residual area | | | Y | Not Estimable |
| 002 | В | $\mathrm{AUC}_{0	ext{-t}}$ | | | N | |
| | | $\mathrm{AUC}_{0	ext{-}\mathrm{inf}}$ | | | N | |
| | | $C_{max}$ | | | Y | Not Estimable |
| | | Residual area | | | Y | Not Estimable |

Treatment A: TRS003, 3 mg/kg IV Infusion Dose; Treatment B: China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose; Treatment C: US Licensed Avastin® (Bevacizumab), 3 mg/kg IV Infusion Dose.

 19-SEP-2018 (Final 1.0)



Zhejiang Teruisi Pharmaceutical Inc.

**Listing 16.2.7-1 Treatment-Emergent Adverse Events** 

| | | | MedDRA® System Organ Class/ | Onset Date and Time/ | | | Action | ı taken | |
|---|---|---|---|---|---|---|---|---|---|
| | | AΕ | MedDRA® Preferred Term/ | Resolution Date and Time | Severity/ | Serious | | | |
| Subject | Treatment | Number | Adverse Event Description | (or Ongoing) | Relationship | (Yes/No) | Study Drug | Other | Outcome |
| 001 | | | SOC 1/ | YYYY-MM-DDTHH:MM/ | Grade 1/ | Yes | | | |
| | | | Preferred Term 1/ | YYYY-MM-DDTHH:MM | Related | | | | |
| | | | DESCRIPTION 1 | | | | | | |
| | | | SOC 2/ | YYYY-MM-DDTHH:MM/ | Grade 2/ | No | | | |
| | | | Preferred Term 2/ | ONGOING | Not Related | | | | |
| | | | DESCRIPTION 2 | | | | | | |

#### Programming Notes:

- 1) SOC and AE Description will be presented in uppercase. The Preferred Term will be presented in "propage". The SAS coding "/~n" between terms will generate the break line.
- 2) The SAS coding "/~n" will generate the break line between dates and between Severity and Relationship.
- 3) If needed, hardcode OUTCOME and ACTIONS in order to introduce break line (~n) between answer elements.
- 4) If medication is ongoing, replace missing resolution date per ONGOING.
- 5) Sort events per Subject, Onset Date/time, Resolution Date/time, SOC and PT.
- 6) For incomplete date display, refer to CDISC SDTM Implementation Guide according to ISO 8601 format.
- 7) Please update' MedDRA® System Organ Class' footnote by keeping only those SOC terms referred in table.

MedDRA®: Medical Dictionary for Regulatory Activities (MedDRA®); MedDRA® Version 21.0.

MedDRA® System Organ Class (SOC): Cardiac disorders (Card); Eye disorders (Eye); Gastrointestinal disorders (Gastr); General disorders and administration site conditions (Genrl); Infections and infestations (Infec); Injury, poisoning and procedural complications (Inj&P); Investigations (Inv); Musculoskeletal and connective tissue disorders (Musc); Nervous system disorders (Nerv); Psychiatric disorders (Psych); Respiratory, thoracic and mediastinal disorders (Resp); Skin and subcutaneous tissue disorders (Skin) Vascular disorders (Vasc).

Treatment A: TRS003, 3 mg/kg IV Infusion Dose; Treatment B: China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose;

Treatment C: US Licensed Avastin® (Bevacizumab), 3 mg/kg IV Infusion Dose.

Note: The list of MedDRA® SOC will be updated according to the AEs observed for the study.

Note: Similar layout will be used for Listing 16.2.7-2, please adapt title and footnotes accordingly.

19-SEP-2018 (Final 1.0) 



Zhejiang Teruisi Pharmaceutical Inc.

**Listing 16.2.8-1 Clinical Laboratory - Biochemistry** 

| | | | Collection Date | | | | |
|---|---|---|---|---|---|---|---|
| Subject | Treatment | Laboratory Visit | and Time | Parameter(unit) | Result | Flag | Normal Range |
| 001 | | | YYYY-MM- | | | Н | XX.X-XX.X |
| | | | DDTHH:MM | | | | |

#### Programming Notes:

- 1) Sort assessments per Subject, Visit/Date and parameters. Sorting for parameter should be as defined in Summary Descriptive Statistics Table.
- 2) For each parameter provide normal range of primary facility and, for gender specific parameters, use the same sorting of gender from demographic table.
- 3) If multiple laboratories involved, display standard and normalised results. Display the ranges in the same way. The SAS coding "/~n" between results or ranges will generate the break line.
  - Take care to use the same precision of both, standard and normalised results/ranges.
- 4) Adapt flag footnote for Urinalysis listing per N: Normal result; A: Abnormal result; H: Above normal range; L: Below normal range.
- 5) Laboratory facilities could be abbreviated with appropriation description on footnote (iHC: inVentiv Health Clinical Laboratory; BML: Biron Medical Laboratory).

H: Above normal range; L: Below normal range; N: Normal Range.

Treatment A: TRS003, 3 mg/kg IV Infusion Dose; Treatment B: China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose;

Treatment C: US Licensed Avastin® (Bevacizumab), 3 mg/kg IV Infusion Dose.

Note: Similar layout will be used for Listings 16.2.8-2, 16.2.8-3 and 16.2.8-6. Please adapt title and footnotes accordingly.

19-SEP-2018 (Final 1.0) 



Zhejiang Teruisi Pharmaceutical Inc.

**Listing 16.2.8-4 Vital Signs Result** 

| Subject | Treatment | Timepoint | Measurement Date and Time | Parameter(unit) | Result |
|---|---|---|---|---|---|
| 001 | A | Screening | YYYY-MM-DDTHH:MM | | |

#### Programming Notes:

1) Sort assessments per Subject, Timepoint/Date and parameter. Parameters for each subject to be sorted as defined in Summary Descriptive Statistics Table.

EOS: End of study; EOI: End of infusion.

Treatment A: TRS003, 3 mg/kg IV Infusion Dose; Treatment B: China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose; Treatment C: US Licensed Avastin<sup>®</sup> (Bevacizumab), 3 mg/kg IV Infusion Dose.

19-SEP-2018 (Final 1.0) 



Zhejiang Teruisi Pharmaceutical Inc.

Listing 16.2.8-5 Electrocardiogram Result

| | 0 | | 8 | | | |
|---|---|---|---|---|---|---|
| Subject | Treatment | Timepoint | Assessment Date and Time | Parameter(unit) | Result/ Interpretation* | Normal range |
| | | | YYYY-MM-DDTHH:MM | | | XX X-XX X |
| | | | | | | 7171.71-7171.71 |

Programming Notes:

1) Sort assessments per Subject, Timepoint/Date and parameter. Parameters for each subject to be sorted as defined in Summary Descriptive Statistics Table.

\*The medical judgement for abnormal ECG interpretation is also presented in this column as CS: Clinically significant or NCS: Not clinically significant.

EOS: End of study; EOI: End of infusion.

Treatment A: TRS003, 3 mg/kg IV Infusion Dose; Treatment B: China-Approved Bevacizumab, 3 mg/kg IV Infusion Dose; Treatment C: US Licensed Avastin<sup>®</sup> (Bevacizumab), 3 mg/kg IV Infusion Dose.

19-SEP-2018 (Final 1.0) 